CLINICAL TRIAL: NCT05441826
Title: A Phase 2 Study of VB119 in Adult Subjects With Steroid-Sensitive Primary Minimal Change Disease (MCD) or Primary Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: Efficacy and Safety of VB119 in Subjects With Minimal Change Disease (MCD) and Focal Segmental Glomerulosclerosis (FSGS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor change
Sponsor: Tenet Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 119-02-02
Record Dates: First submitted 2022-06-07; First posted 2022-07-01 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Minimal Change Disease; Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VB119 (Experimental): VB119 100 or 200mg IV doses administered 4 times
  Interventions: Drug: VB119

INTERVENTIONS:
Drug: VB119 — Humanized, immunoglobin (Ig) G1 monoclonal antibody (mAb) to be administered as intravenous infusion at multiple timepoints during the study.

SUMMARY:
Phase 2, multi-center, proof-of-concept study to evaluate the safety and efficacy of VB119 on the maintenance of remission and duration of response in adults with primary MCD or primary FSGS who previously responded to steroid therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Is ≥ 18 years of age at the time of informed consent;
2. Kidney biopsy-proven diagnosis of primary MCD or primary FSGS within the past 10 years. Subjects with kidney biopsy-proven diagnosis of primary MCD or primary FSGS greater than 10 years and less than 20 years prior to Screening who meet all other eligibility criteria may be enrolled after discussion with the Medical Monitor
3. History of steroid-sensitive MCD or FSGS, defined as having achieved complete remission of proteinuria (reduction of proteinuria to <0.5 g/g UPCR) after use of corticosteroids;
4. Has experienced meaningful proteinuria in the last 2 years prior to Screening, defined as UPCR >2.0 g/g, after attempted or completed tapering of steroids and/or CNIs that occurs within 6 months of the attempt or completion of tapering;
5. Currently on prednisone regimen at time of Screening and anticipated to be tapered to a stable dose of prednisone of no more than 20 mg/day for at least 14 days prior to Day 1
6. Has systolic blood pressure (BP) <160 mmHg or diastolic BP <100 mmHg after 5 minutes of rest at Screening;
7. Is willing and able to provide written informed consent prior to Screening;
8. Female subjects of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before the Screening Visit) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone in the postmenopausal range at Screening, based on the central laboratory's ranges;
9. Female subjects of childbearing potential (ie, ovulating, premenopausal, or not surgically sterile) and all male subjects must use a medically accepted, highly effective contraceptive regimen during their participation in the study and for 125 days (4 months) after the last administration of study drug.
10. Male subjects must agree to abstain from sperm donation through 125 days (4 months) after administration of the last dose of study drug.

Exclusion Criteria:

1. Has an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 at Screening utilizing the Chronic Kidney DiseaseEpidemiology Collaboration formula confirmed by the central laboratory;
2. Has an absolute neutrophil count <1.5 x 10/L;
3. Has a white blood cell count <3.0 x 10/L;
4. Has secondary causes of MCD or FSGS (eg, malignancy, hepatitis B or C, human immunodeficiency virus [HIV], systemic lupus erythematosus [SLE], or other autoimmune diseases [eg, thyroiditis], drug-induced);
5. Has a diagnosis or history of SLE (including non renal disease);
6. Has type 1 or 2 diabetes mellitus;
7. Has an acute, chronic, or latent infection, including tuberculosis, hepatitis, HIV, or chronic urinary tract infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects in remission at End of Treatment | Day 274
  Efficacy
Incidence of serious adverse events (SAEs) | through Day 420
  Safety and Tolerability
Incidence of treatment-emergent adverse events (TEAEs) | through Day 420
  Safety and Tolerability
Incidence of adverse events of special interest (AESIs) | through Day 420
  Safety and Tolerability

SECONDARY OUTCOMES:
Change in UPCR | Multiple timepoints from Day 1 to Day 337
  Efficacy
Change in eGFR | Multiple timepoints from Screening to Day 337
  Efficacy
Proportion of subjects that are recurrence-free | From Day 1 to Day 337
  Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Keenan, Study Chair — ValenzaBio, Inc.
Locations (1):
- Clinical Research Site, Albany, New York, United States